CLINICAL TRIAL: NCT06034756
Title: Temporomandibular Joint Problems, Head Posture, Tongue Strength and Endurance and Core Stabilization With University Students
Brief Title: Temporomandibular Joint Problems and Core Stabilization
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Other Study IDs: 2022-18
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Temporomandibular Joint Disorders; Core Stability
Keywords: temporomandibular disorders; core stability; head posture; tongue strength
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TMJ dysfunction — Fonseca's Anamnestic Questionnaire (FAQ) was used for TMJ dysfunction. The diagnostic accuracy of the FAQ was found to be high in identifying pain-related and intra-articular TMDs, and the cut-off point was set as 25 points. A score of 25 and above was accepted as the presence of TMD.
Other: Maximum pain-free mouth opening (MMO) — The maximum pain-free mouth opening was recorded using a 15 cm ruler
Other: Forward head posture — Forward head posture was evaluated by CVA using a goniometer. CVA was measured in degrees as the angle between the horizontal plane, the seventh cervical vertebra and the ear hole
Other: Tongue strength and endurance — Tongue strength and endurance were evaluated with IOPI (Medical LLC, Redmond, WA), which has been clinically validated and reliable
Other: Static endurance evaluation of the trunk muscles — The Trunk Flexors Endurance Test and the Biering Sorenson Test were used. These static tests are measurements targeting the local core muscles.
Other: Dynamic endurance evaluation of the core muscles — The Sit-ups and the Modified Push-ups Tests were used. These dynamic tests are measurements targeting the global core muscles.

SUMMARY:
This study aimed to investigate the relationship between temporomandibular joint problems, head posture, tongue strength, and endurance with core stabilization.

DETAILED DESCRIPTION:
This cross-sectional study was conducted on university students aged 18-31 between September 2022 and February 2023. In the evaluation of the students were used that the Fonseca's Anamnestic Questionnaire for temporomandibular joint dysfunction, Research Diagnostic Criteria for Temporomandibular Disorders Examination Form for maximum pain-free mouth opening, presence of sound in temporomandibular joint movements, and palpation parameters of temporomandibular joint and surrounding muscles, Craniovertebral Angle for forward head posture, and Iowa Oral Performance Instrument for tongue strength and endurance. In addition, the Trunk Flexor Endurance Test and Biering Sorenson Test were used for static endurance of the core muscles, and Sit-ups Test and Modified Push-ups Test were used for dynamic endurance of the core muscles.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18 and 31 who agreed to participate in the study
* signed the Informed Consent Form were included.

Exclusion Criteria:

* having a non-reducible disc problem,
* having surgery related to spine, abdomen and/or TMJ problem,
* history of trauma, cancer,
* presence of neurological problems, congenital anomaly, musculoskeletal problems, systemic disease, facial paralysis,
* receiving any treatment related to the spine and TMJ in less than six months.

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
TMJ dysfunction | September 2022- February 2023
  Fonseca's Anamnestic Questionnaire (FAQ) was used for TMJ dysfunction. The FAQ has a multi-factor evaluation structure. The questionnaire consists of ten questions about pain in TMJ, head, and joints, with answer options of "No, Sometimes and Yes." A score of 25 and above was accepted as the presence of TMD.
Maximum pain-free mouth opening (MMO) | September 2022- February 2023
  The maximum pain-free mouth opening was recorded using a 15 cm ruler
Forward head posture | September 2022- February 2023
  Forward head posture was evaluated by CVA using a goniometer.
Tongue strength and endurance | September 2022- February 2023
  Tongue strength and endurance were evaluated with IOPI (Medical LLC, Redmond, WA), which has been clinically validated and reliable
Static endurance evaluation of the trunk muscles | September 2022- February 2023
  The Trunk Flexors Endurance Test and the Biering Sorenson Test were used. These static tests are measurements targeting the local core muscles. The time the individuals maintained their position was recorded in seconds (sec) using a stopwatch.
Dynamic endurance evaluation of the core muscles: | September 2022- February 2023
  The Sit-ups and the Modified Push-ups Tests were used. These dynamic tests are measurements targeting the global core muscles. The number of times the individuals could perform the movement for 30 sec was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided